CLINICAL TRIAL: NCT00671671
Title: A Phase 1, Non- Randomized, Open Label, Sequential Group, Multicenter Study To Evaluate The Antiviral Activity Of Multiple Doses Of A Small Molecule Direct Antiviral Agent In Chronically Infected Hepatitis C Subjects.
Brief Title: Phase 1 Study To Evaluate Antiviral Activity Of Small Molecule Direct Antiviral Agent At Multiple Doses In Subjects With Chronically Infected Hepatitis C Virus.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A8121006
Record Dates: First submitted 2008-04-25; First posted 2008-05-05 (Estimated); Results first posted 2014-01-14 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2013-11

CONDITIONS: Hepatitis, Chronic; Hepatitis C Virus
MeSH Terms: conditions — Hepatitis, Chronic; Hepatitis C | interventions — filibuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort B (Experimental)
  Interventions: Drug: Small Molecule Agent (PF-868554)
- Cohort A (Experimental): Dose study drug in subjects who have previously failed to respond to interferon based therapies
  Interventions: Drug: Small Molecule Agent (PF-868554)

INTERVENTIONS:
Drug: Small Molecule Agent (PF-868554) — Study drug will be administered 700mg BID in the fed state for three days.
  Arms: Cohort B
Drug: Small Molecule Agent (PF-868554) — Study drug will be given 450mg BID for a duration of 10 days.
  Arms: Cohort A

SUMMARY:
Phase 1 study in HVC (Hepatitis C Virus) infected subjects to determine pharmacokinetics, safety and efficacy in subjects with no or inadequate response to prior treatment.

ELIGIBILITY:
Inclusion Criteria:

HCV Positive With HCV RNA>100,000 iu/ml Genotype 1; COHORT A- non responders or partial

Exclusion Criteria:

HIV HBV co-infection Decompensated liver disease Liver disease due to causes other than HCV, AFP>200ng/ml

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Gainesville, Florida, United States

REFERENCES:
- [Derived] Wagner F, Thompson R, Kantaridis C, Simpson P, Troke PJ, Jagannatha S, Neelakantan S, Purohit VS, Hammond JL. Antiviral activity of the hepatitis C virus polymerase inhibitor filibuvir in genotype 1-infected patients. Hepatology. 2011 Jul;54(1):50-9. doi: 10.1002/hep.24342. PMID 21488067
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8121006&StudyName=Phase%201%20Study%20To%20Evaluate%20Antiviral%20Activity%20Of%20Small%20Molecule%20Direct%20Antiviral%20Agent%20At%20Multiple%20Doses%20In%20Subjects%20With%20Chronically%20I

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-00868554 450 mg (Cohort A): Participants who had a history of unsuccessful treatment for hepatitis C virus (HCV) with an interferon-alpha (IFN-alpha) regimen (with or without ribavirin [RBV]) due to lack of response or relapse, received PF-00868554 450 milligram (mg) tablet orally twice daily, every 12 hours from Day 1 morning dose to Day 10 morning dose in a fasted state.
- PF-00868554 700 mg (Cohort B): Participants who did not receive any prior treatment for HCV with an IFN-alpha regimen (with or without RBV) or who discontinued from an IFN-alpha regimen (with or without RBV) after less than or equal to (<=) 2 weeks of treatment due to tolerability issues or other reasons, received PF-00868554 700 mg tablet orally twice daily, every 12 hours from Day 1 morning dose to Day 3 evening dose in a fed state.
Period: Overall Study
Arm/Group | PF-00868554 450 mg (Cohort A) | PF-00868554 700 mg (Cohort B)
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-00868554 450 mg (Cohort A) | PF-00868554 700 mg (Cohort B) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Customized [Number; unit: participants]
  18 to 44 years | 1 | 2 | 3
  45 to 64 years | 9 | 7 | 16
  greater than or equal to (>=) 65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Plasma Log10 Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) at Day 11 (Cohort A): Full Analysis Set
Description: Plasma HCV RNA levels were quantified using the Abbott RealTime HCV assay (lower limit of quantification [LLOQ] = 12 international unit per milliliter [IU/mL]). Baseline value calculated as an average of screening, Day 0 and Day 1 (0 hour) measurements. Change from baseline in plasma log10 HCV RNA was calculated for all participants after the last day of dosing (Day 11 for Cohort A).
Time Frame: Baseline, Day 11
Population: Full Analysis Set (FAS) included all randomized participants who took at least 1 dose of study medication and had both baseline and at least 1 valid post-baseline endpoint measurements for HCV viral load.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | PF-00868554 450 mg (Cohort A)
Number analyzed (Participants) | 10
log10 IU/mL
  Baseline | 6.11 (0.449)
  Change at Day 11 | -0.45 (0.439)

2. Primary Outcome: Change From Baseline in Plasma Log10 Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) at Day 11 (Cohort A): Modified Analysis Set
Description: Plasma HCV RNA levels were quantified using the Abbott RealTime HCV assay (LLOQ = 12 IU/mL). Baseline value calculated as an average of screening, Day 0 and Day 1 (0 hour) measurements. Change from baseline in plasma log10 HCV RNA was calculated for all participants after the last day of dosing (Day 11 for Cohort A).
Time Frame: Baseline, Day 11
Population: Modified Analysis Set (MAS): a subset of FAS which included all participants who had received complete dosage in the corresponding treatment regimen.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | PF-00868554 450 mg (Cohort A)
Number analyzed (Participants) | 10
log10 IU/mL
  Baseline | 6.11 (0.449)
  Change at Day 11 | -0.45 (0.439)

3. Primary Outcome: Change From Baseline in Plasma Log10 Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) at Day 4 (Cohort B): Full Analysis Set
Description: Plasma HCV RNA levels were quantified using the Abbott RealTime HCV assay (LLOQ = 12 IU/mL). Baseline value calculated as an average of screening, Day 0 and Day 1 (0 hour) measurements. Change from baseline in plasma log10 HCV RNA was calculated for all participants after the last day of dosing (Day 4 for Cohort B).
Time Frame: Baseline, Day 4
Population: FAS included all randomized participants who took at least 1 dose of study medication and had both baseline and at least 1 valid post-baseline endpoint measurements for HCV viral load.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | PF-00868554 700 mg (Cohort B)
Number analyzed (Participants) | 10
log10 IU/mL
  Baseline | 6.39 (0.455)
  Change at Day 4 | -2.15 (0.252)

4. Primary Outcome: Change From Baseline in Plasma Log10 Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) at Day 4 (Cohort B): Modified Analysis Set
Description: Plasma HCV RNA levels were quantified using the Abbott RealTime HCV assay (LLOQ = 12 IU/mL). Baseline value calculated as the average of screening, Day 0 and Day 1 (0 hour) measurements. Change from baseline in plasma log10 HCV RNA was calculated for all participants after the last day of dosing (Day 4 for Cohort B).
Time Frame: Baseline, Day 4
Population: MAS: a subset of FAS which included all participants who had received complete dosage in the corresponding treatment regimen.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | PF-00868554 700 mg (Cohort B)
Number analyzed (Participants) | 10
log10 IU/mL
  Baseline | 6.39 (0.455)
  Change at Day 4 | -2.15 (0.252)

5. Primary Outcome: Change From Baseline in Plasma Log10 Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) at Nadir: Full Analysis Set
Description: Plasma HCV RNA levels were quantified using the Abbott RealTime HCV assay (LLOQ = 12 IU/mL). Change from baseline in plasma Log10 HCV RNA at nadir signified the maximum change observed during the study.
Time Frame: Baseline, Nadir (lowest HCV RNA level), assessed up to Day 11 for Cohort A and Day 4 for Cohort B
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | PF-00868554 450 mg (Cohort A) | PF-00868554 700 mg (Cohort B)
Number analyzed (Participants) | 10 | 10
log10 IU/mL | -2.2 (0.23) | -2.3 (0.34)

6. Primary Outcome: Change From Baseline in Plasma Log10 Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) at Nadir: Modified Analysis Set
Description: as for outcome 5
Time Frame: Baseline, Nadir (lowest HCV RNA level), assessed up to Day 11 for Cohort A and Day 4 for Cohort B
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | PF-00868554 450 mg (Cohort A) | PF-00868554 700 mg (Cohort B)
Number analyzed (Participants) | 10 | 10
log10 IU/mL | -2.2 (0.23) | -2.3 (0.34)

7. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau)
Description: Area under the concentration curve from time 0 to end of dosing interval (AUCtau), where dosing interval was 12 hours. AUCtau was evaluated at first dose on Day 1 for Cohort A and B, and at last dose for Cohort A (Day 10) and Cohort B (Day 3).
Time Frame: Predose, 0.5, 1, 2, 6, 8, 12 hours (hrs) postdose on Day 1 for Cohort A and B, pre-evening dose, 0.5, 1, 2, 4, 6, 8, 12 hrs post-evening dose on Day 3 for Cohort B, predose, 0.5, 1, 2, 4, 8, 12 hrs postdose on Day 10 for Cohort A
Population: Per Protocol (PP) analysis set included all participants who took PF-00866554 and had sufficient plasma concentration data to facilitate calculation of the pharmacokinetic (PK) parameters. Here 'n' signifies those participants who were evaluable for this measure at specified time points for each arm, respectively.
Measure: Geometric Mean (Standard Deviation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | PF-00868554 450 mg (Cohort A) | PF-00868554 700 mg (Cohort B)
Number analyzed (Participants) | 10 | 10
nanogram*hour/milliliter (ng*hr/mL)
  Day 1 (n=10, 10) | 140275.9 (38990.36) | 198506.9 (79422.27)
  Day 3 for Cohort B (n=0, 10) | NA (NA) — Data was not collected for this arm at given time point as per planned analysis. | 291172.4 (184959.54)
  Day 10 for Cohort A (n=10, 0) | 139239.7 (94286.82) | NA (NA) — Data was not collected for this arm at given time point as per planned analysis.

8. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the serum concentration time-curve from zero to the last measured concentration (AUClast). AUClast was evaluated at first dose on Day 1 for Cohort A and B, and at last dose for Cohort A (Day 10) and Cohort B (Day 3).
Time Frame: Predose, 0.5, 1, 2, 6, 8, 12, 14 hrs postdose on Day 1 for Cohort A, B, pre-morning dose, pre-evening dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 48 hrs post-evening dose on Day 3 for Cohort B, predose,0.5, 1, 2, 4, 8, 12, 24, 48 hrs postdose on Day 10 for Cohort A
Population: PP analysis set. 'N' (number of participants analyzed) = participants evaluable for this measure. 'n' = participants evaluable for this measure at specified time points for each arm, respectively. Given the sampling schedule on Day 1 and Day 10 for 450 mg dose in Cohort A, AUClast data was not considered meaningful and hence were not analyzed.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PF-00868554 450 mg (Cohort A) | PF-00868554 700 mg (Cohort B)
Number analyzed (Participants) | 0 | 10
ng*hr/mL
  Day 1 (n=0, 10) |  | 239697.9 (93463.98)
  Day 3 for Cohort B (n=0, 10) |  | 344075.5 (248444.34)

9. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)]
Description: AUC (0 - ∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞). AUC (0 - ∞) was evaluated at last dose for Cohort A (Day 10) and Cohort B (Day 3).
Time Frame: Pre-morning dose, pre-evening dose, 0.5, 1, 2, 4, 6, 8, 12, 24, 48 hrs post-evening dose on Day 3 for Cohort B, predose,0.5, 1, 2, 4, 8, 12, 24, 48 hrs postdose on Day 10 for Cohort A
Population: PP analysis set. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. Results are reported for Cohort B at Day 3. Due to differences in sampling schedules between Cohort A and B, AUC (0 - ∞) data was not considered meaningful and hence were not analyzed on Day 10 for Cohort A.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PF-00868554 450 mg (Cohort A) | PF-00868554 700 mg (Cohort B)
Number analyzed (Participants) | 0 | 10
ng*hr/mL |  | 346170.1 (250370.33)

10. Secondary Outcome: Plasma Concentration at The End of Dosing Interval (Ctau)
Description: Ctau was evaluated at first dose on Day 1 for Cohort A and B, and at last dose for Cohort A (Day 10) and Cohort B (Day 3).
Time Frame: as for outcome 7
Population: PP analysis set. Here 'n' signifies those participants who were evaluable for this measure at specified time points for each arm, respectively. The Ctau on Day 1 was not necessary for interpretation of the PK data and hence was not analyzed.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-00868554 450 mg (Cohort A) | PF-00868554 700 mg (Cohort B)
Number analyzed (Participants) | 10 | 10
ng/mL
  Day 3 for Cohort B (n=0, 10) | NA (NA) — Data was not collected for this arm at given time point as per planned analysis. | 6572.0 (9550.56)
  Day 10 for Cohort A (n=10, 0) | 1435.2 (3065.84) | NA (NA) — Data was not collected for this arm at given time point as per planned analysis.

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Cmax was evaluated at first dose on Day 1 for Cohort A and B, and at last dose for Cohort A (Day 10) and Cohort B (Day 3).
Time Frame: as for outcome 8
Population: PP analysis set included all participants who took PF-00866554 and had sufficient plasma concentration data to facilitate calculation of the PK parameters. Here 'n' signifies those participants who were evaluable for this measure at specified time points for each arm, respectively.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-00868554 450 mg (Cohort A) | PF-00868554 700 mg (Cohort B)
Number analyzed (Participants) | 10 | 10
ng/mL
  Day 1 (n=10, 10) | 44688.1 (13542.30) | 38734.5 (14464.27)
  Day 3 for Cohort B (n=0, 10) | NA (NA) — Data was not collected for this arm at given time point as per planned analysis. | 50274.1 (22297.74)
  Day 10 for Cohort A (n=10, 0) | 42859.7 (16697.78) | NA (NA) — Data was not collected for this arm at given time point as per planned analysis.

12. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Description: Tmax was evaluated at first dose on Day 1 for Cohort A and B, and at last dose for Cohort A (Day 10) and Cohort B (Day 3).
Time Frame: as for outcome 8
Population: as for outcome 11
Measure: Median (Full Range); unit: hours
Arm/Group | PF-00868554 450 mg (Cohort A) | PF-00868554 700 mg (Cohort B)
Number analyzed (Participants) | 10 | 10
hours
  Day 1 (n=10, 10) | 0.750 [0.50 to 2.00] | 2.000 [1.00 to 2.00]
  Day 3 for Cohort B (n=0, 10) | NA [NA to NA] — Data was not collected for this arm at given time point as per planned analysis. | 2.000 [1.00 to 4.00]
  Day 10 for Cohort A (n=10, 0) | 1.000 [0.50 to 2.00] | NA [NA to NA] — Data was not collected for this arm at given time point as per planned analysis.

13. Secondary Outcome: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half. Half-life was evaluated at last dose for Cohort A (Day 10) and Cohort B (Day 3).
Time Frame: as for outcome 9
Population: PP analysis set. 'N' (number of participants analyzed) = participants evaluable for this measure. Results are reported for Cohort B at Day 3. Due to limited sampling, time interval over which plasma concentrations were measured after final dose was too short relative to projected t1/2. Therefore, t1/2 estimates were not calculated on Day 10.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PF-00868554 450 mg (Cohort A) | PF-00868554 700 mg (Cohort B)
Number analyzed (Participants) | 0 | 10
hours |  | 7.468 (1.3235)

ADVERSE EVENTS:
Arm/Group | PF-00868554 450 mg (Cohort A) | PF-00868554 700 mg (Cohort B)
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 10/10 | 7/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-00868554 450 mg (Cohort A) (N=10) | PF-00868554 700 mg (Cohort B) (N=10)
Ear pain (Ear and labyrinth disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 4 | 1
Eructation (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Stomach discomfort (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Pain (General disorders) | 1 | 2
Rhinitis (Infections and infestations) | 0 | 1
Tinea pedis (Infections and infestations) | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 4 | 3
Haematuria (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.